CLINICAL TRIAL: NCT02024191
Title: The Role of Glutamine for Preventing Oxaliplatin-Induced Peripheral Neuropathy in Colorectal Cancer Patients. Randomized Trial
Brief Title: The Role of Glutamine for Preventing Oxaliplatin-Induced Peripheral Neuropathy
Acronym: GELUPO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ozan Yazici, MD, Ankara Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 031
Record Dates: First submitted 2013-12-25; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Peripheral Neuropathy
Keywords: glutamine; oxaliplatin; peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Glutamine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glutamine (Experimental): The patient group had 3x10 gr daily glutamine during first 4 cycles of mFOLFOX6 regimen.
  Interventions: Dietary Supplement: Glutamine
- Observation (No Intervention): The group who had only mFOLFOX6 regimen, no additional intervention for neuropathy prophylaxis..

INTERVENTIONS:
Dietary Supplement: Glutamine
  Other Names: Resource Glutamine 3x10 gr per day
  Arms: Glutamine

SUMMARY:
Oxaliplatin is a chemotherapeutic agent, which is generally used in treatment of colorectal cancer. The dose limiting side effect of oxaliplatin is neurotoxicity. In this study we aimed to determine whether glutamine has role in prevention of oxaliplatin induced neuropathy.

DETAILED DESCRIPTION:
Our study population includes the colorectal cancer patient who is going to have mFOLFOX6 (modified, Folinic acid 400 mg/m2 1 day, oxaliplatin 85 mg/m2 1 day, 5-fluorouracil l 400 mg/m2 bolus 2400 mg/m2 continuous infusion 48 hours) regimen. We randomly assigned the patients into two groups. We administered glutamine at dose of 3x10 gr/day to one patient group concomitantly with mFOLFOX6 regimen and other group had no additional intervention. We performed questionnaire, neurological examination and EMG (Electromyography) before and after 4th cycle of mFOLFOX6 regimen in both patient groups. We planned to compare the neurological signs, symptoms and EMG action potentials between mFOLFOX6+Glutamine and only mFOLFOX6 group. We aimed to search the role of glutamine as a prophylactic agent against oxaliplatin induced neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 - 65 years
* Operated and non operated colorectal cancer patients
* Patient administering mFOLFOX 6 ( Folinic acid 400 mg/m2 1 day, oxaliplatin 85 mg/m2 1 day, 5-fluorouracil 400 mg/m2 bolus 2400 mg/m2 continuous infusion 48 hours)

Exclusion Criteria:

* Patients who had chemotherapy in last 6 months
* Diabetes Mellitus
* Sensorimotor polyneuropathy
* Anemia

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-01 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Electromyography parameters | 4 months interval
  Electromyography action potential values will be compared between two patient groups.

SECONDARY OUTCOMES:
Neurological signs and symptoms | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Numune Education and Research Hospital, Ankara, Turkey (Türkiye)